CLINICAL TRIAL: NCT05838352
Title: The Effect of Physiotherapy and Nutrition Services Provided by Telerehabilitation Method on the Physical, Nutrition and Psychological Conditions of Children With Autism and Their Families
Brief Title: Multidisciplinary Telerehabilitation Practices in Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tele_autism
Record Dates: First submitted 2022-12-09; First posted 2023-05-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Physiotherapy and Rehabilitation; Nutrition; Autism Spectrum Disorder; Telerehabilitation
Keywords: Physiotherapy and Rehabilitation; Nutrition; Autism Spectrum Disorder; Telerehabilitation; Multidisciplinary
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Resistance Training; Nutrition Assessment; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (TRG) (Experimental): The group given physical activity and nutrition counseling for 2 months through telerehabilitation.
  Interventions: Other: telerehabilitation exercise
- Conventional Rehabilitation Group (CRG) (Active Comparator): The group who received conventional treatment and had no intervention, only pretest measurements
  Interventions: Other: Control Group

INTERVENTIONS:
Other: telerehabilitation exercise — The telerehabilitation program is as follows; Respiratory exercises: Chest, diaphragmatic breathing and lower basal breathing exercises will be performed with 10 repetitions.Resistance exercises: Strengthening exercises will be performed on the major muscle groups of the upper and lower extremities, using medium-hardness resistance exercise band. During the exercises, the patient's fatigue and dyspnea levels will be questioned using the Borg scale, and breaks will be given when necessary. Exercises 1st-3rd weeks with 10 repetitions; 15 repetitions in weeks 4-6; In the 7th and 8th weeks, it will be done as 2 sets of 10 repetitions.Posture exercises: Basic posture exercises will be explained. Tabletop movements will be taught in clear, various positions that concern the spine, scapula and pelvis.Gait training: In line with the data obtained from the 6-minute walking test, gait training will be given on flat ground at 60% workload (land-based walking).
  Other Names: Exercise program; Physical Activity Education; Nutrition Education
  Arms: Telerehabilitation Group (TRG)
Other: Control Group — The surveys in the outcome measures section will be applied once as a pre-test. Children in both groups will receive conventional institutional rehabilitation in the rehabilitation center. Children in the conventional rehabilitation group, which is the control group, will only be included in the supervised program. This group will not receive a telerehabilitation program.
  Arms: Conventional Rehabilitation Group (CRG)

SUMMARY:
The study, titled The Effect of Physiotherapy and Nutrition Services Provided by Telerehabilitation Methods on the Physical, Nutritional and Psychological Conditions of Children with Autism and Their Families, aimed to evaluate the effects of physiotherapy and nutrition education to be given to the participants. Participants were children with autism spectrum disorder and parents of children with autism spectrum disorder. There will be surveys that researchers will ask participants to answer. Parent telerehabilitation group participants via smartphone video conferencing; Researchers involved in this project; A physiotherapist and a physiotherapist senior physiotherapy intern will send 1 session of online simultaneous exercise training to the parent telerehabilitation group participants, then an exercise video containing the exercises and brochures will be sent and the parent telerehabilitation group participants will be asked to do the exercises 3 days a week. Participants will be asked to keep an exercise diary and the status of the diaries will be monitored once a week. Additionally, the concepts of physical activity and recreational activity in autism will be explained to the participants. Again, via smartphone video conferencing, the researchers participating in this project; 3 different nutrition trainings will be given by 1 dietitian and 1 senior dietitian trainee within the scope of basic nutrition and nutrition-health information at 15-day intervals. Waist, hip and height measurements of autistic child participants will be measured with a tape measure, and their body weight will be measured with a scale. The study will last 2 months.

DETAILED DESCRIPTION:
There are studies in the literature to investigate physical activity and nutrition in the diagnosis of Autism Spectrum Disorder (ASD). This project will be a multidisciplinary and comprehensive study conducted on children with ASD and their parents with the participation of a physiotherapist and dietitian in Turkey. It will contribute to the literature as it is a randomized controlled study that evaluates primary school age (6-11) children with autism from a multidisciplinary perspective in terms of physiotherapy and nutrition and provides physical activity and nutrition education to the family. In this study, there are two groups: telerehabilitation group and control group; There are 4 participant types: telerehabilitation parent, telerehabilitation child, control parent, control child. The surveys for both groups are in the form of pre-test and post-test. Quality of life, activity participation and recreational activity levels of children with autism will be measured. In line with these measurements, recreational activities that will guide telerehabilitation parent participants in ASD will be explained and consultancy will be given on their implementation. For all participating parents; Quality of life, functional status and stress levels will be evaluated. As a result of these evaluations, breathing, resistance and posture exercises and walking training will be given and the effectiveness of these trainings will be evaluated. In this training, the current approach, telerehabilitation, will be used. Telerehabilitation is a cost-effective, easy-to-access alternative to traditional treatment options.

In the literature, attention is drawn to nutritional problems such as food rejection, food selectivity, and obesity in children with ASD. Adequate and balanced nutrition is very important for children's mental and physical health, growth and development. For this purpose, it was aimed to raise awareness of the participants about nutrition. In the study, the nutritional status, food consumption frequency and food selectivity/rejection of children with ASD will be determined. Anthropometric measurements such as height, weight, upper middle arm circumference (UMAC), and body mass index (BMI) will be taken and evaluated according to the children's age and gender. The nutritional knowledge level of all participating parents will be measured at the beginning, and the knowledge level at the end of the study will be determined by providing nutrition education during the study.

The training will be given simultaneously, using technological devices, and the training will be transferred as a video later so that parents can easily access it.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* 6-11 years old child
* Have an approved medical diagnosis for Asperger's syndrome, autism, or a specific developmental disorder (DSM 5), by the standards set in the Diagnostic and Statistical Manual of Mental Disorders, fifth edition
* Children with mild to moderate autism according to the childhood autism rating scale
* Not having received physical activity and nutrition counseling before
* Children with normal orally fed and functioning gastrointestinal tract

Exclusion Criteria:

* Having any serious condition (such as orthopedic or any acute) for which it is contraindicated to the viewer of recreational entertainment programs
* Recent (less than 4 weeks) children on any psychotropic medication
* Those who have high-intensity activity according to the International Physical Activity Questionnaire (IPAQ)
* Children with chewing and swallowing difficulties
* You can enter as a child suitable for children.
* Children with diagnosed nutritional problems (absorption disorder, metabolic structure)
* have Gastroenterol patients suitable for medical intervention or bowel segments,
* Leukemia or other cancers,
* Hypothyroidism or other chronic conditions that can grow and turn into energy
* Acute myocarditis, active endocarditis, control eg missed heart probe, tachyarrhythmia, bradyarrhythmia, hypertrophic cardiomyopathy

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure for Children (WeeFIM) | Change from baseline WeeFIM score at 6 weeks
  Functional Independence measure for children (WeeFIM) is an adaptation of the Functional Independence Measure (FIM) developed for adults. It is a useful, short and comprehensive measurement tool that detects the developmental, educational and social functional limitations of children with Cerebral Palsy and other developmental disorders. WeeFIM consists of 18 items in 6 areas The scores that can be obtained from the scale are between 18 and 126. The higher the score, the higher the child's independence. A higher score indicates positive improvement.
Quality of Life Questionnaire in Autism | Change from baseline Quality of Life Questionnaire in Autism score at 6 weeks
  It has been divided into two subsections (A and B). Part A contains 28 questions that measure how parents perceive their quality of life. Part B contains 20 questions that assess parents' perceptions of how much of a problem their child's autism-specific difficulties are for them. In the five-point Likert-type assessment measure, in which they evaluate how problematic these situations are for the parents, five are scored as 'It was not a problem for me at all', while one is scored as 'It was a lot of trouble for me'. The score that can be obtained from the scale is between 48-240. A high score indicates an improved quality of life.
Cornell musculoskeletal discomfort questionnaire | Change from baseline Cornell musculoskeletal discomfort questionnaire score at 6 weeks
  The questionnaire surveyed the frequency and severity of pain or discomfort in 11 different body regions (neck, shoulder, back, upper arm, wrist, forearm, wrist, hip, upper leg, knee, and lower leg) during the work period in the last week. assessing its impact on performance. For each body region, the weighted score of that body region is calculated by multiplying the ratings marked from the areas of frequency, severity, and effect on work performance. Scores for each region range from 0 to 90. A high score indicates that the region has a pain and disability.
Beck Depression Inventory | Change from baseline Beck Depression Inventory score at 6 weeks
  It is used to objectively determine the level of depression exhibited by individuals. Beck Depression Inventory includes 21 categories of depressive symptoms. Each of these categories consists of 4 items for self-assessment and is graded between 0 and 3 points.
6 minutes walking test | Change from baseline 6 minute walking distance at 6 weeks
  The 6-minute walk test measures the distance the patient can walk quickly on a flat, hard surface in a period of 6 minutes. It evaluates the integrated responses of all systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. The vital signs of the participants were taken before and after the test. The 6 minute walk test (6MWT) built in a 30 m-long straight corridor. The patient was asked to walk as much as they could, and the distance walked was recorded in meters.
Evaluation of Participation in Activities | Change from baseline Evaluation of Participation in Activities at 6 weeks
  In the study, with the form the investigators created to evaluate the participation of children with special needs in leisure activities, the demographic characteristics of the children, their educational status, the economic status of their families, the type and reason for their disability were asked to the families, which activities they wanted to do and what they did, the situations that prevented them from participating in the activities and the assistive tools they used were asked to the children. evaluated.
Evaluation of Family Role in Activity Participation | Change from baseline Evaluation of Family Role in Activity Participation at 6 weeks
  A form was created that included the questions of who decides the activities that the children will do, whether the families control them during the activity, whether the children are willing to participate in the activity and whether they can express the activity they participate in, to what extent the families approve of their children's ideas and to what extent they encourage their children to participate in the activities. the role was evaluated.
Childhood Autism Rating Scale | Change from baseline Childhood Autism Rating Scale score at 6 weeks
  The Childhood Autism Rating Scale can be applied to children of all age groups starting from the preschool period. It is a 15-item scale that evaluates behaviors in 14 areas that are generally affected by serious problems in autism and a general impression category of autism. Each question has a rating of 1-4. It means mild autism between 15 and 29 points, moderate autism between 30 and 36 points and severe autism between 37 and 60 points.
Food Consumption Frequency Questionnaire | Change from baseline Food Consumption Frequency Questionnaire score at 6 weeks
  In order to determine the food consumption status of children with autism, it was applied to parents of children with an autism spectrum disorder. The questionnaire separates 5 food groups and includes the foods belonging to each food group under these groups. The frequency of food consumption was determined by the answer given to the words written opposite the food: Every day, 2-3 times a week, once a week, 2-3 times a month, once a month, or never.
Autism Meal Behavior Brief Scale | Change from baseline Autism Meal Behavior Brief Scale score at 6 weeks
  The scale aims to evaluate the nutritional problems observed in individuals with autism and intellectual disability. It consists of three subscales and 18 items: food refusal, limitation in food variety, and behavioral characteristics related to autism. Food refusal (5-25 points) subscale consists of 5 items, food diversity restriction subscale (8-40 points) consists of 8 items and autism-related behavioral characteristics subscale (5-25 points) consists of 5 items. The scale is in a five-point Likert type and the 3rd, 9th, 10th and 15th items are scored in reverse. A high total score from the scale indicates the severity of nutritional problems, it means negative.
Nutrition Knowledge Level Scales | Change from baseline Nutrition Knowledge Level Scales score at 6 weeks
  It is a scale that measures the level of nutrition knowledge. It consists of two parts. first part; It contains 20 questions containing basic nutrition and nutrition-health information. The second part is the part where food preference is questioned, which consists of 12 questions. The first part that questions the basic knowledge level is between 0-80 points, and the higher the score, the higher the level of knowledge. The second section questioning food preference is between 0-48 points, and the higher the score, the better the food choice.

SECONDARY OUTCOMES:
Body mass index calculation | Change from baseline Body mass index at 6 weeks
  After determining the height and weight, it will be calculated with the kilogram/square meter formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided